CLINICAL TRIAL: NCT05690594
Title: Evaluation of Long-term Outcomes on Urinary Continence, Fecal Continence, Sexuality and Quality of Life of Patients Treated for Bladder Exstrophy by Questionnaires.
Brief Title: Long-term Outcomes of Patients Treated for Bladder Exstrophy by Questionnaires.
Acronym: QUALEXSTRO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1072
Record Dates: First submitted 2023-01-06; First posted 2023-01-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Bladder Exstrophy
Keywords: Bladder exstrophy; Quality of life; Urinary continence; Fecal continence
MeSH Terms: conditions — Bladder Exstrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self or straight administered questionnaire — Self or straight administered questionnaire with 5 parts:
  * General questionnaire (to collect socio-demographic data)
  * ICIQ score to evaluate urinary continence
  * FLQI score to evaluate fecal continence
  * FSFI score to evaluate sexuality in women or IIEF-5 score to evaluate sexuality in men
  * SF-12 score to evaluate quality of life The questionnaire will be sent to patients by email and/or mail. Patients will be able to either complete the questionnaire alone and return it to the primary investigator, or to request a telephone interview to help them to complete the questionnaire. The questionnaire is administered only once and the estimated response time to the questionnaire is between 30 minutes and one hour.

SUMMARY:
The bladder exstrophy epispadias complex (BEEC) is a rare spectrum of congenital conditions due to abnormal development of the cloacal membrane. Of these conditions, bladder exstrophy (BE) represent a mild form and requires several complex surgical corrections to gain access to a urinary and fecal acceptable continence and a normal sexual function at adulthood. Despite the surgeries, patients may suffer, in the long term, from functional impairments (incontinence, sexuality disorders) which can impact severely their quality of life. However, only a few studies investigate long term issues of bladder exstrophy patients, with heterogenous population and small samples.

The department of pediatric surgery of the Hospices Civils of Lyon is an expert center in the management of patients born with bladder exstrophy. At adulthood, departments of adult urology continue the follow-up and treat residual complications. Thus, a large cohort of adults and adolescents' patients with bladder exstrophy is currently followed at our institution.

Therefore, the aim of this study is to evaluate urinary continence, fecal continence, sexuality and quality of life among a large cohort of patients treated for bladder exstrophy, using questionnaires.

All patients over 15 years old and treated for bladder exstrophy at our institution are included in the study. Exclusion's criteria are : patients treated for epispadias or cloacal exstrophy, patients initially treated of their bladder exstrophy abroad with no access to the surgical report, patients under a guardianship measure. All included patients are contacted by e-mail or phone to answer the questionnaire. The purpose of statistical analysis is to evaluate the average score in each field of investigation:

* Mean ICIQ score for urinary continence
* Mean FLQI score for fecal continence
* Mean FSFI score for sexuality in women
* Mean IIEF-5 score for sexuality in men
* Mean SF-12 score for quality of life, in comparison of mean SF-12 score in general French population based on literature

Secondary objectives are to assess the impact of different surgical strategies used for bladder exstrophy reparation on urinary continence, fecal continence, sexuality and quality of life ; to describe the population from a sociological point of view (level of study, profession, marital status) and to describe the population reproductive status (pregnancy, delivery modalities, paternity and maternity status, use of medically assisted procreation).

ELIGIBILITY:
Inclusion Criteria:

* Patients born with bladder exstrophy or cloacal exstrophy
* Aged 15 and over at time of enrolment
* Treated at the Hospices Civils of Lyon

Exclusion Criteria:

* patients treated for epispadias
* patients initially treated of their bladder exstrophy abroad with no access to the surgical report
* patients under a guardianship measure
* deceased patients

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population is selected on the database of the hospital. All patients over 15 years old and treated for bladder exstrophy or cloacal exstrophy at our institution are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Assessment of average score of ICIQ score for urinary continence | At inclusion
  The study is descriptive, and the purpose is to evaluate the average score in each field of investigation:
  - Mean ICIQ score for urinary continence
Assessment of FLQI score for fecal continence | At inclusion
  - Mean FLQI score for fecal continence
Assessment of FSFI score and IIEF-5 score for sexuality in women and men | At inclusion
  * Mean FSFI score for sexuality in women
  * Mean IIEF-5 score for sexuality in men
Assessment of SF-12 score for quality of life | At inclusion
  - Mean SF-12 score for quality of life, in comparison of mean SF-12 score in general French population based on literature.
  Data on the average SF-12 score for the French population are available in the Gandek et al study, which validated the French version of the score in 1998.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Femme mère et enfant, Bron